CLINICAL TRIAL: NCT03467802
Title: Porcine Collagen Matrix With and Without Enamel Matrix Derivative for the Treatment of Gingival Recession Defects
Brief Title: Collagen Matrix With and Without Enamel Matrix Derivative
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: WRNMMC-2017-0123
Record Dates: First submitted 2018-03-01; First posted 2018-03-16 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-04

CONDITIONS: Gingival Recession
Keywords: Gingival Recession; Enamel Matrix Derivative; Porcine Collagen Matrix
MeSH Terms: conditions — Gingival Recession | interventions — enamel matrix proteins

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Biological: enamel matrix derivative — Enamel matrix derivative (EMD), sold under the brand name Emdogain®, is an amelogenin derivative of embryonal porcine enamel and is FDA approved for application to root surfaces to treat recession defects. Amelogenins comprise the majority of the proteins in EMD while others such as tuftelin, ameloblastin and amelin make up the remainder. EMD is thought to mimic the role of proteins crucial to cementogenesis and root development, which may promote new gingival attachment to exposed roots. The properties of EMD may favor early healing of the soft tissue and stimulate angiogenesis.
  Other Names: Emdogain®
Device: Porcine collagen matrix — Mucograft® is a bi-layered grafting material composed of Type I and III collagen. It is derived from veterinary certified pigs, sterilized by gamma irradiation and has a low antigenicity in conjunction with good biocompatibility. The material is approximately 2.5-5mm thick and is indicated for root coverage, increasing keratinized tissue, covering of implants placed immediately and alveolar ridge reconstruction. A compact outer layer contributes to protection, structure and allows for better control during suturing; while the inner layer is thick, porous and spongy in nature, providing a suitable environment for early vascularization and promotion of cellular in-growth.
  Other Names: Mucograft®

SUMMARY:
The purpose of this prospective, double-blinded, randomized, split-mouth study is to compare the effectiveness of a porcine collagen matrix (CM) and coronally advanced flap (CAF) with or without the addition of enamel matrix derivative (EMD) in the treatment of Miller Class I, II, or predictable class III recession defects. One defect will receive CM + CAF + EMD (Experimental), while the other will receive CM + CAF (Control) alone. The treatment of 60 similarly sized Miller class I, II, or predictable class III recession defects on single-rooted teeth in 30 subjects using CM + CAF + EMD or CM + CAF alone will be evaluated. The subjects will be in good health, non-smokers, periodontally healthy with good oral hygiene and have no contraindications to periodontal surgery. Paired, similar sized defects on single-rooted teeth will be in the same subject and measure within 2mm of each other. One defect will be randomly assigned as the test group using CM + CAF + EMD, and the other as the control group using only CM + CAF. Clinical measurements will be made using a UNC-15 periodontal probe by calibrated, board certified periodontists and will include: probing depth (PD), clinical attachment level (CAL), vertical recession (RD), and width of keratinized tissue (KT). Percent root coverage (%RC) will be calculated. The measurements will be used to evaluate surgical outcome. Surgical outcome will also be assessed using stone models. All measurements will be taken at baseline (on the day of the surgery) and 3 and 6 months post-surgery for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Patient will remain in the Capital region for at least 6 months following the surgical procedure for follow up appointments
* Patient must be otherwise periodontally healthy
* Patient must be systemically healthy (ASA class I or II)
* Patient must have no contraindications to periodontal surgery
* Patient must have demonstrated good oral hygiene (plaque index <1 according to Silness and Löe)
* Paired Miller Class I, II or predictable III recession defects
* Bilateral, facial defects on single-rooted teeth

Exclusion Criteria:

* Self-reported history of smoking within previous 6 months
* Does not meet any of the preceding criteria
* Female patients who are pregnant or nursing
* Antibiotic medications taken within the last 6 months
* History of mucogingival surgery at the sites of interest
* Poor plaque control (>25% of sites)
* Those with clinically significant systemic disease, which may affect healing (i.e. uncontrolled diabetes or bone metabolic disease)
* Allergy to chlorhexidine gluconate (Peridex)
* Does not sign study consent or HIPAA forms
* Bleeding complications (e.g. hemophilia)
* Warfarin therapy
* History of osteoporosis or taking bisphosphonate medications
* History of radiation therapy in the head and neck area
* Mobile teeth beyond physiologic mobility
* Facial restorations at the site to be treated
* Recession defects that will require more than one 15x20mm Mucograft (per side)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants must meet health eligibility requirements and not have any conditions that will exclude them from the study (see exclusion criteria below). Females of reproductive age will be asked to submit urine samples for pregnancy testing prior to surgery. Urine HCG tests will be conducted in the Department of Periodontics in accordance with WRNNMC Bethesda Point of Care Testing Procedures. Pregnant females will be excluded from this study in accordance with standard of care (periodontal surgery is routinely deferred during pregnancy).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in gingival recession using conventional measurements | Baseline to 6 months
  Change in gingival recession measurements from baseline to 6 months
Change in root coverage using digital analysis | Baseline to 6 months
  Assessment of surgical outcome by optically scanning stone models captured at baseline to 6 months post-surgery. The digital files will be aligned using global registration and GR recorded by measuring the distance from cemento-enamel junction to the height of the marginal gingiva using computer software. % RC will be calculated by comparing GR at the various times.
Change in Probing Depths | Baseline to 6 months
  Change in Probing Depthmeasurements from baseline to 6 months
Change in Clinical Attachment Levels | Baseline to 6 months
  Change in Clinical Attachment Levels measurements from baseline to 6 months
Change in Keratinized Tissue | Baseline to 6 months
  Change in Keratinized Tissue measurements from baseline to 6 months

SECONDARY OUTCOMES:
Comparison of digital vs. conventional measurement | Baseline to 6 months
  Compare conventional and digital change in gingival recession to assess the two modalities treatment outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed NMMC, Bethesda, Maryland, United States